CLINICAL TRIAL: NCT00799838
Title: Local, Phase IV, Multicenter, Double-blind, Randomized, Parallel, With Two Treatment Arms, Placebo-controlled Study to Evaluate the Reduction of Inflammatory Symptoms in the Treatment of Bacterial Pharyngitis With Ketoprofen and Amoxicillin in Pediatric Patients.
Brief Title: Evaluation of Inflammatory Symptoms Reduction With Amoxicillin + Ketoprofen in Acute Pharyngeal Tonsillitis in Pediatric Patients
Acronym: DROPS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment challenges despite several attenpts to increase enrollment
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KETOP_L_03102; 2014-004002-15 (EudraCT Number)
Record Dates: First submitted 2008-11-28; First posted 2008-12-01 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-03

CONDITIONS: Pharyngotonsillitis
MeSH Terms: interventions — Ketoprofen; Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketoprofen + Amoxicillin (Experimental): Ketoprofen + Amoxicillin for 3 days, then Amoxicillin alone for 7 days
  Interventions: Drug: Ketoprofen; Drug: Amoxicillin
- Amoxicillin (Placebo Comparator): Placebo (for ketoprofen) + Amoxicillin for 3 days, then Amoxicillin alone for 7 days
  Interventions: Drug: Placebo (for Ketoprofen); Drug: Amoxicillin

INTERVENTIONS:
Drug: Ketoprofen — Formulation: oral solution 20mg/mL
  Route of administration: oral
  Dose regimen: 1 drop/Kg for children aged between 4 to 6 years old or 25 drops for children from 7 to 11 years old administered t.i.d
  Arms: Ketoprofen + Amoxicillin
Drug: Placebo (for Ketoprofen) — Formulation: oral solution
  Route of administration: oral
  Dose regimen: 1 drop/Kg for children aged between 4 to 6 years old or 25 drops for children from 7 to 11 years old administered t.i.d
  Arms: Amoxicillin
Drug: Amoxicillin — Formulation: suspension 125mg/5 mL
  Route of administration: oral
  Dose regimen: 20-40mg/Kg/day administered t.i.d

SUMMARY:
The purpose of this study is to evaluate the inflammatory symptoms and signs (hyperemia, edema and pain) reduction after 24 hours of treatment with ketoprofen drops when associated to amoxicillin.

DETAILED DESCRIPTION:
The total duration of the study period per patient is 10 ± 1 day

ELIGIBILITY:
Inclusion Criteria:

* Quick-test positive for Streptococcus pyogenes;
* Indication for treatment with amoxicillin according to labeling and physician's clinical evaluation;
* Pain (for swallowing) evaluated by Wong Baker Faces Pain scale with at least grade 3;
* Presence of at least two of the follow symptoms:

  * Hyperemia and edema evaluated with at least 2 out of 4 crosses
  * Fever in the previous 48 hours
  * Cervical adenomegaly
  * Tonsilla with erythema or erythema and white exsudate.

Exclusion Criteria:

* History of cardiovascular, gastrointestinal, metabolic or psychiatric conditions;
* History and laboratorial confirmation of hematologic, hepatic or renal disorders;
* Use of nonsteroidal antiinflammatory drugs (NSAID) during the last 3 weeks and gastroesophageal reflux during the last 6 months;
* Use of analgesic or anti inflammatory medication (except Paracetamol) in the previous 12 hours;
* History of allergy or hypersensitivity to amoxicillin and/ or ketoprofen.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2008-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with reduction of inflammatory signs and symptoms after 24 hours of treatment | 24 hours

SECONDARY OUTCOMES:
Number of patients with reduction of inflammatory signs and symptoms after 72 hours of treatment | 72 hours
Number of patients with reduction of inflammatory signs and symptoms with no use of rescue medication | 24 hours and 72 hours
Number of patients who used rescue medication after randomization. | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil